CLINICAL TRIAL: NCT04132518
Title: A Randomized, Multi-center, Evaluator-blinded, No-treatment Controlled Study to Evaluate the Effectiveness and Safety of Sculptra for Correction of Midface Volume Deficit and/or Midface Contour Deficiency
Brief Title: Sculptra for Correction of Midface Volume Deficit and/or Midface Contour Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43CHSA1803
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-01

CONDITIONS: Midface Volume Deficit
Keywords: PLLA; Midface Volume Deficit

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Sculptra (Experimental): Participants in Group A will receive up to 4 injections of Sculptra from Day 1 with 5 (±1) weeks (at least 4 weeks) intervals and will be followed up for 24 months.
  Interventions: Device: Sculptra
- Group B: Sculptra (Experimental): Participants in Group B will receive up to 4 injections of Sculptra from Day 1 with 5 (±1) weeks (at least 4 weeks) intervals and will be followed up for 24 months.
  Interventions: Device: Sculptra
- Group B: Control (No Intervention): Participants in Group B will not receive any treatment and participants will be followed up for 12 months.

INTERVENTIONS:
Device: Sculptra — Initial injection and optional 3 injections with Sculptra in Midface.
  Arms: Group A: Sculptra; Group B: Sculptra

SUMMARY:
This is a randomized, evaluator-blinded, no-treatment controlled study in participants with Midface Volume Deficit and/or Midface Contour Deficiency.

DETAILED DESCRIPTION:
For Group A, after screening, eligible participants will be treated from day 1 and followed up for 24 months. The purpose of Group A was to confirm investigator's use of correct injection technique.

For Group B, the study includes two phases as follows:

Main study phase: It is randomized, evaluator-blinded and no-treatment controlled. After screening, all eligible participants will be randomized either to the Treatment Group or the Control Group in a 2:1 ratio. All the participants will be followed up for 12 months.

Extension study phase: After the main study phase, the Treatment Group will be followed up for additional 12 months.

Each subject assigned to Group A and Treatment Group will receive up to 4 injection sessions with 5(±1) weeks intervals.

Participants assigned to the Control Group will not receive treatment during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent to participate in the study.
2. Men or women aged 18 years of age or older of Chinese origin.
3. Participants seeking augmentation therapy for the midface.
4. MMVS score of 2, 3 or 4 on each side of the face as assessed by the blinded evaluator.

Exclusion Criteria:

1. Known/previous allergy or hypersensitivity to any of the constituents of the product.
2. Known/previous allergy or hypersensitivity to local anaesthetics, e.g. lidocaine or other amide-type anaesthetics.
3. History of severe or multiple allergies, such as anaphylaxis.
4. Previous tissue revitalization treatment with laser or light, mesotherapy, radiofrequency, ultrasound, cryotherapy, chemical peeling or dermabrasion in the area to be treated within 6 months before treatment.
5. Previous surgery (including aesthetic facial surgical therapy or liposuction), piercing or tattoo in the area to be treated.
6. Previous tissue augmentation therapy or contouring with any permanent (non-biodegradable) or semi-permanent filler, autologous fat, lifting threads or permanent implant in the area to be treated.
7. Other condition preventing the subject from entering the study in the Investigator's opinion, e.g. participants not likely to avoid other facial cosmetic treatments, participants anticipated to be unreliable, unavailable or incapable of understanding the study assessments or having unrealistic expectations of the treatment result.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2021-07-18 (Actual); Study Completion 2022-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galderma, Study Director — Galderma R&D
Locations (6):
- China (6):
  - Galderma research site 3, Beijing
  - Galderma research site 4, Beijing
  - Galderma research site 5, Chengdu
  - Galderma research site 2, Guangzhou
  - Galderma research site 6, Hangzhou
  - Galderma research site 1, Shanghai

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 centers in China from 12 November 2019 to 18 July 2022.
Pre-assignment Details: A total of 16 participants were enrolled into Group A and 189 participants were enrolled into Group B. Out of 189 participants in Group B, 126 participants randomized in treatment group and 63 participants in control group or no treatment group.
Groups:
- Group A: Sculptra: Participants in Group A received up to 4 injections of Sculptra from Day 1 with 5 (±1) weeks (at least 4 weeks) intervals and were followed up for 24 months.
- Group B: Sculptra: Participants in Group B received up to 4 injections of Sculptra from Day 1 with 5 (±1) weeks (at least 4 weeks) intervals and were followed up for 24 months.
- Group B: Control: Participants in Group B did not receive any treatment and followed up for 12 months.
Period: Overall Study
Arm/Group | Group A: Sculptra | Group B: Sculptra | Group B: Control
Started | 16 | 126 | 63
Treated | 16 | 124 | 0
Completed | 16 | 117 | 62
Not Completed | 0 | 9 | 1
Not completed — Prematurely withdrawn from the study | 0 | 9 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants in Group B who were treated with Sculptra or randomized to no-treatment group and participant in Group A who were treated with Sculptra.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Sculptra | Group B: Sculptra | Group B: Control | Total
Number analyzed (Participants) | 16 | 124 | 63 | 203
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (9.6) | 41.3 (10.2) | 40.5 (10.7) | 40.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 116 | 54 | 183
  Male | 3 | 8 | 9 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese Han | 16 | 116 | 60 | 192
  Other | 0 | 8 | 3 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  China | 16 | 124 | 63 | 203

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 1 Point Improvement From Baseline on the Medicis Midface Volume Scale (MMVS) as Measured by the Blinded Evaluator at Month 12
Description: MMVS is a 4-grade scale that assesses the fullness of the midface from Fairly Full (1) to Substantial Loss of Fullness (4) as described below. The blinded evaluator and treating investigator rated the participant's right and left midface for severity of volume deficiency using the MMVS at all applicable study visits. A one grade decrease in score from baseline was defined as a treatment success/improvement, meaning that lower score means a better outcome.
  1. Fairly full midface
  2. Mild loss of fullness in midface area
  3. Moderate loss of fullness with slight hollowing below malar prominence
  4. Substantial loss of fullness in the midface area, clearly apparent hollowing below malar prominence
Time Frame: Baseline, Month 12
Population: FAS included all participants in Group B who were treated with Sculptra or randomized to no-treatment group and participant in Group A who were treated with Sculptra.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group A: Sculptra | Group B: Sculptra | Group B: Control
Number analyzed (Participants) | 16 | 124 | 63
Percentage of participants | 68.8 [41.3 to 89.0] | 69.4 [60.4 to 77.3] | 1.6 [0.0 to 8.5]

2. Secondary Outcome: Percentage of Participants With 1 Point Improvement From Baseline on the MMVS as Measured by the Blinded Evaluator
Description: as for outcome 1
Time Frame: Treatment group: Baseline, Months 6, 9, 18 and 24; Control group: Baseline, Months 6 and 9
Population: Full analysis set (FAS) included all participants in Group B who were treated with Sculptra or randomized to no-treatment group and participant in Group A who were treated with Sculptra. "Here, 'Overall number of participants analyzed' signifies participants who were evaluable for this outcome measure and number analyzed signifies who were evaluable at the given timepoints.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group A: Sculptra | Group B: Sculptra | Group B: Control
Number analyzed (Participants) | 16 | 124 | 62
Percentage of participants
  At Month 6 | 81.3 [54.4 to 96.0] | 68.5 [59.6 to 76.6] | 3.2 [0.4 to 11.2]
  At Month 9: number analyzed (Participants) | 16 | 122 | 62
  At Month 9 | 62.5 [35.4 to 84.8] | 68.0 [59.0 to 76.2] | 3.2 [0.4 to 11.2]
  At Month 18: number analyzed (Participants) | 16 | 118 | 0
  At Month 18 | 68.8 [41.3 to 89.0] | 59.3 [49.9 to 68.3] |
  At Month 24: number analyzed (Participants) | 16 | 117 | 0
  At Month 24 | 56.3 [29.9 to 80.2] | 59.0 [49.5 to 68.0] |

3. Secondary Outcome: Percentage of Participants With 1 Point Improvement From Baseline on the MMVS as Measured by the Treating Investigator
Description: as for outcome 1
Time Frame: Treatment group: Baseline, Months 6, 9, 12, 18 and 24; Control group: Baseline, Months 6, 9 and 12
Population: FAS included all participants in Group B who were treated with Sculptra or randomized to no-treatment group and participant in Group A who were treated with Sculptra. "Here, 'Overall number of participants analyzed' signifies participants who were evaluable for this outcome measure and number analyzed signifies who were evaluable at the given timepoints.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group A: Sculptra | Group B: Sculptra | Group B: Control
Number analyzed (Participants) | 16 | 124 | 62
Percentage of participants
  At Month 6 | 93.8 [69.8 to 99.8] | 81.5 [73.5 to 87.9] | 6.5 [1.8 to 15.7]
  At Month 9: number analyzed (Participants) | 16 | 122 | 62
  At Month 9 | 93.8 [69.8 to 99.8] | 80.3 [72.2 to 87.0] | 4.8 [1.0 to 13.5]
  At Month 12: number analyzed (Participants) | 16 | 122 | 62
  At Month 12 | 87.5 [61.7 to 98.4] | 82.8 [74.9 to 89.0] | 6.5 [1.8 to 15.7]
  At Month 18: number analyzed (Participants) | 16 | 118 | 0
  At Month 18 | 87.5 [61.7 to 98.4] | 72.0 [63.0 to 79.9] |
  At Month 24: number analyzed (Participants) | 16 | 117 | 0
  At Month 24 | 62.5 [35.4 to 84.8] | 73.5 [64.5 to 81.2] |

4. Secondary Outcome: Total Volume Change From Baseline Over Time of the Right and Left Midface Areas
Description: Total volume change from baseline over time (both sides of the face combined) was calculated by a digital 3D image analysis.
Time Frame: Treatment group: Baseline, Months 6, 9, 12, 18 and 24; Control group: Baseline, Months 6, 9 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | Group A: Sculptra | Group B: Sculptra | Group B: Control
Number analyzed (Participants) | 16 | 124 | 62
milliliter (mL)
  Month 6: number analyzed (Participants) | 16 | 124 | 61
  Month 6 | 2.15 (1.19) | 1.96 (1.03) | 0.15 (0.82)
  Month 9: number analyzed (Participants) | 16 | 122 | 62
  Month 9 | 2.63 (1.59) | 2.46 (1.26) | 0.13 (0.72)
  Month 12: number analyzed (Participants) | 16 | 122 | 62
  Month 12 | 2.74 (1.72) | 2.81 (1.28) | 0.20 (0.83)
  Month 18: number analyzed (Participants) | 16 | 114 | 0
  Month 18 | 3.27 (1.71) | 2.94 (1.35) |
  Month 24: number analyzed (Participants) | 16 | 115 | 0
  Month 24 | 3.10 (1.38) | 3.00 (1.48) |

5. Secondary Outcome: Percentage of Responders According to the Global Aesthetic Improvement Scale (GAIS) on Both Sides of the Face Combined as Assessed by the Treating Investigator
Description: The 5-graded GAIS was used to live assess the aesthetic improvement of the midface fullness of both sides of the participant's face as compared to photographs taken before treatment. Each midface side was rated separately. Rating and its Description:1. Very much improved (Optimal cosmetic result for the implant in this participant), 2. Much improved (Marked improvement in appearance from the original condition),3. Improved (Obvious improvement in appearance from the original condition), 4. No change (The appearance is essentially the same as original condition), 5. Worse (The appearance is worse than the original condition). Responders are those with a rating of at least improved. Participants with a GAIS rating of 'Very much improved', 'Much improved', or 'Improved' are defined as responders. Percentage of responders," according to the GAIS on both sides of the face combined, as assessed by the Treating Investigator was reported.
Time Frame: Treatment group: Months 6, 9, 12, 18 and 24; Control group: Months 6, 9 and 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | Group A: Sculptra | Group B: Sculptra | Group B: Control
Number analyzed (Participants) | 16 | 124 | 62
Percentage of responders
  Month 6 | 100.0 [79.4 to 100.0] | 97.6 [93.1 to 99.5] | 3.2 [0.4 to 11.2]
  Month 9: number analyzed (Participants) | 16 | 122 | 62
  Month 9 | 93.8 [69.8 to 99.8] | 98.4 [94.2 to 99.8] | 1.6 [0.0 to 8.7]
  Months 12: number analyzed (Participants) | 16 | 122 | 62
  Months 12 | 100.0 [79.4 to 100.0] | 96.7 [91.8 to 99.1] | 1.6 [0.0 to 8.7]
  Month 18: number analyzed (Participants) | 16 | 118 | 0
  Month 18 | 100.0 [79.4 to 100.0] | 98.3 [94.0 to 99.8] |
  Month 24: number analyzed (Participants) | 16 | 117 | 0
  Month 24 | 93.8 [69.8 to 99.8] | 95.7 [90.3 to 98.6] |

6. Secondary Outcome: Percentage of Responders According to the GAIS on Both Sides of the Face Combined as Assessed by the Participant
Description: The 5-graded GAIS was used to live assess the aesthetic improvement of the midface fullness of both sides of the participant's face as compared to photographs taken before treatment. Each midface side was rated separately. Rating and its Description: 1. Very much improved (Optimal cosmetic result for the implant in this participant), 2. Much improved (Marked improvement in appearance from the original condition),3. Improved (Obvious improvement in appearance from the original condition), 4. No change (The appearance is essentially the same as original condition), 5. Worse (The appearance is worse than the original condition). Responders are those with a rating of at least improved. Participants with a GAIS rating of 'Very much improved', 'Much improved', or 'Improved' are defined as responders. Percentage of responders," according to the GAIS on both sides of the face combined, as assessed by the Participant was reported.
Time Frame: Treatment group: Months 6, 9, 12, 18 and 24; Control group: Months 6, 9 and 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | Group A: Sculptra | Group B: Sculptra | Group B: Control
Number analyzed (Participants) | 16 | 124 | 62
Percentage of responders
  Month 6 | 100.0 [79.4 to 100.0] | 96.0 [90.8 to 98.7] | 1.6 [0.0 to 8.7]
  Month 9: number analyzed (Participants) | 16 | 122 | 62
  Month 9 | 93.8 [69.8 to 99.8] | 95.9 [90.7 to 98.7] | 0.0 [0.0 to 0.1]
  Month 12: number analyzed (Participants) | 16 | 122 | 62
  Month 12 | 100.0 [79.4 to 100.0] | 95.1 [89.6 to 98.2] | 0.0 [0.0 to 0.1]
  Month 18: number analyzed (Participants) | 16 | 118 | 0
  Month 18 | 100.0 [79.4 to 100.0] | 92.4 [86.0 to 96.5] |
  Month 24: number analyzed (Participants) | 16 | 117 | 0
  Month 24 | 100.0 [79.4 to 100.0] | 89.7 [82.8 to 94.6] |

7. Secondary Outcome: Percentage of Participants Agreeing That Their Cheek Volume Deficit and/or Contour Deficiency Was Improved by the Treatment
Description: The subject's satisfaction with the procedure was assessed using a Subject Satisfaction Questionnaire. Question 1 was a YES or NO question pertaining to satisfaction with study treatment: Do you think your Cheek Volume deficit and/or Contour Deficiency has been improved with the treatment?
Time Frame: Treatment group: Months 6, 9, 12, 18 and 24
Population: FAS included all participants in Group B who were treated with Sculptra or randomized to no-treatment group and participant in Group A who were treated with Sculptra. "Here, number analyzed signifies who were evaluable at the given timepoints. Data was planned to be analyzed and collected only for treatment group.
Measure: Number; unit: percentage of participants
Arm/Group | Group A: Sculptra | Group B: Sculptra
Number analyzed (Participants) | 16 | 124
percentage of participants
  Month 6 | 93.8 | 93.5
  Month 9: number analyzed (Participants) | 16 | 122
  Month 9 | 93.8 | 95.9
  Month 12: number analyzed (Participants) | 16 | 122
  Month 12 | 93.8 | 94.3
  Month 18: number analyzed (Participants) | 16 | 118
  Month 18 | 100.0 | 92.4
  Month 24: number analyzed (Participants) | 16 | 117
  Month 24 | 100.0 | 94.0

8. Secondary Outcome: Percentage of Participants Agreeing That Overall Result of the Treatment Looks Natural
Description: The subject's satisfaction with the procedure was assessed using a Subject Satisfaction Questionnaire. Question 2 was a YES or NO question pertaining to naturalness of the study treatment: Do you think that the overall result of the treatment looks natural?
Time Frame: Treatment group: Months 6, 9, 12, 18 and 24
Population: FAS included all participants in Group B who were treated with Sculptra or randomized to no-treatment group and participant in Group A who were treated with Sculptra. "Here, 'Overall number of participants analyzed' signifies participants who were evaluable for this outcome measure and number analyzed signifies who were evaluable at the given timepoints. Data was planned to be analyzed and collected only for treatment group.
Measure: Number; unit: percentage of participants
Arm/Group | Group A: Sculptra | Group B: Sculptra
Number analyzed (Participants) | 16 | 124
percentage of participants
  Month 6 | 100.0 | 98.4
  Month 9: number analyzed (Participants) | 16 | 122
  Month 9 | 100.0 | 97.5
  Month 12: number analyzed (Participants) | 16 | 122
  Month 12 | 93.8 | 98.4
  Month 18: number analyzed (Participants) | 16 | 118
  Month 18 | 100.0 | 97.5
  Month 24: number analyzed (Participants) | 16 | 117
  Month 24 | 93.8 | 97.4

9. Secondary Outcome: Percentage of Participants Agreeing That the Treatment Met or Surpassed Their Expectations to the Study Treatment
Description: The subject's satisfaction with the procedure was assessed using a Subject Satisfaction Questionnaire. Question 3 was answered on a 4-grade scale: Would you say that the study treatment: Surpass your expectations/Meet your expectations/ Do Meet your expectations/You did not have any specific expectations before the injections?
Time Frame: Treatment group: Months 6, 9, 12, 18 and 24
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Group A: Sculptra | Group B: Sculptra
Number analyzed (Participants) | 16 | 124
percentage of participants
  Month 6: Meet your expectations | 62.5 | 69.4
  Month 6: Surpass your expectations | 31.3 | 12.9
  Month 9: Meet your expectations: number analyzed (Participants) | 16 | 122
  Month 9: Meet your expectations | 62.5 | 75.4
  Month 9: Surpass your expectations | 25.0 | 9.8
  Month 12: Meet your expectations: number analyzed (Participants) | 16 | 122
  Month 12: Meet your expectations | 62.5 | 73.8
  Month 12: Surpass your expectations | 31.3 | 13.9
  Month 18: Meet your expectations: number analyzed (Participants) | 16 | 118
  Month 18: Meet your expectations | 50.0 | 67.8
  Month 18: Surpass your expectations | 43.8 | 17.8
  Month 24: Meet your expectations: number analyzed (Participants) | 16 | 117
  Month 24: Meet your expectations | 43.8 | 67.5
  Month 24: Surpass your expectations | 43.8 | 20.5

10. Secondary Outcome: Percentage of Participants Agreeing That Treatment Brings More "Youth/Beauty/Harmony/Symmetrical Appearance/Pep/Liveliness/Freshened Look/Self-esteem/Confidence"
Description: The subject's satisfaction with the procedure was assessed using a Subject Satisfaction Questionnaire. Question 4 was a yes or no question: Do you think that the treatment brings you more: Youth/Beauty/Harmony/Symmetrical appearance/Pep/Liveliness/Freshened look/Self-esteem/confidence.
Time Frame: Treatment group: Months 6, 9, 12, 18 and 24
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Group A: Sculptra | Group B: Sculptra
Number analyzed (Participants) | 16 | 124
percentage of participants
  Month 6 : Youth | 87.5 | 58.1
  Month 6 : Beauty | 31.3 | 29.8
  Month 6 : Harmony | 50.0 | 41.1
  Month 6 : Symmetrical appearance | 43.8 | 24.2
  Month 6 : Pep/Liveliness /Freshened look | 12.5 | 44.4
  Month 6 : Selfesteem/ confidence | 31.3 | 25.8
  Month 9: Youth: number analyzed (Participants) | 16 | 122
  Month 9: Youth | 62.5 | 55.7
  Month 9 : Beauty: number analyzed (Participants) | 16 | 122
  Month 9 : Beauty | 43.8 | 34.4
  Month 9 : Harmony: number analyzed (Participants) | 16 | 122
  Month 9 : Harmony | 50.0 | 50.0
  Month 9: Symmetrical appearance: number analyzed (Participants) | 16 | 122
  Month 9: Symmetrical appearance | 25.0 | 27.0
  Month 9: Pep/Liveliness /Freshened look: number analyzed (Participants) | 16 | 122
  Month 9: Pep/Liveliness /Freshened look | 56.3 | 41.8
  Month 9 : Selfesteem/ confidence: number analyzed (Participants) | 16 | 122
  Month 9 : Selfesteem/ confidence | 18.8 | 22.1
  Month 12: Youth: number analyzed (Participants) | 16 | 122
  Month 12: Youth | 100.0 | 60.7
  Month 12 : Beauty: number analyzed (Participants) | 16 | 122
  Month 12 : Beauty | 37.5 | 28.7
  Month 12 : Harmony: number analyzed (Participants) | 16 | 122
  Month 12 : Harmony | 43.8 | 47.5
  Month 12: Symmetrical appearance: number analyzed (Participants) | 16 | 122
  Month 12: Symmetrical appearance | 31.3 | 32.0
  Month 12 : Pep/Liveliness /Freshened look: number analyzed (Participants) | 16 | 122
  Month 12 : Pep/Liveliness /Freshened look | 50.0 | 36.9
  Month 12: Selfesteem/ confidence: number analyzed (Participants) | 16 | 122
  Month 12: Selfesteem/ confidence | 37.5 | 27.9
  Month 18: Youth: number analyzed (Participants) | 16 | 118
  Month 18: Youth | 68.8 | 61.9
  Month 18 : Beauty: number analyzed (Participants) | 16 | 118
  Month 18 : Beauty | 37.5 | 29.7
  Month 18 : Harmony: number analyzed (Participants) | 16 | 118
  Month 18 : Harmony | 50.0 | 48.3
  Month 18 : Symmetrical appearance: number analyzed (Participants) | 16 | 118
  Month 18 : Symmetrical appearance | 25.0 | 22.0
  Month 18: Pep/Liveliness /Freshened look: number analyzed (Participants) | 16 | 118
  Month 18: Pep/Liveliness /Freshened look | 68.8 | 39.8
  Month 18: Selfesteem/ confidence: number analyzed (Participants) | 16 | 118
  Month 18: Selfesteem/ confidence | 31.3 | 28.8
  Month 24 : Youth: number analyzed (Participants) | 16 | 117
  Month 24 : Youth | 75.0 | 59.0
  Month 24 : Beauty: number analyzed (Participants) | 16 | 117
  Month 24 : Beauty | 43.8 | 38.5
  Month 24 : Harmony: number analyzed (Participants) | 16 | 117
  Month 24 : Harmony | 43.8 | 50.4
  Month 24 : Symmetrical appearance: number analyzed (Participants) | 16 | 117
  Month 24 : Symmetrical appearance | 25.0 | 31.6
  Month 24 : Pep/Liveliness /Freshened look: number analyzed (Participants) | 16 | 117
  Month 24 : Pep/Liveliness /Freshened look | 37.5 | 44.4
  Month 24 : Selfesteem/ confidence: number analyzed (Participants) | 16 | 117
  Month 24 : Selfesteem/ confidence | 37.5 | 26.5

11. Secondary Outcome: Percentage of Participants Agreeing That They Feel More Attractive by the Treatment
Description: The subject's satisfaction with the procedure was assessed using a Subject Satisfaction Questionnaire. Question 5 was a yes or no question: Would you say that you feel more attractive?
Time Frame: Treatment group: Months 6, 9, 12, 18 and 24
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Group A: Sculptra | Group B: Sculptra
Number analyzed (Participants) | 16 | 124
percentage of participants
  Month 6: Yes | 100.0 | 80.6
  Month 9: Yes: number analyzed (Participants) | 16 | 122
  Month 9: Yes | 93.8 | 85.2
  Month 12 : Yes: number analyzed (Participants) | 16 | 122
  Month 12 : Yes | 93.8 | 86.9
  Month 18: Yes: number analyzed (Participants) | 16 | 118
  Month 18: Yes | 93.8 | 84.7
  Month 24 : Yes: number analyzed (Participants) | 16 | 117
  Month 24 : Yes | 87.5 | 88.9

12. Secondary Outcome: Percentage of Participants Agreeing That They Feel Better by the Treatment
Description: The subject's satisfaction with the procedure was assessed using a Subject Satisfaction Questionnaire. Question 6 was answered on a 5-grade scale: How do you feel about yourself since the treatment was performed? Very much better / Much better / Somewhat better / The same / Worse. Percentage of participants who responded Very much better / Much better / Somewhat better were reported in this outcome measure.
Time Frame: Treatment group: Months 6, 9, 12, 18 and 24
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Group A: Sculptra | Group B: Sculptra
Number analyzed (Participants) | 16 | 124
percentage of participants
  Month 6 : Very much better | 50.0 | 15.3
  Month 6 : Much better | 12.5 | 47.6
  Month 6 : Somewhat better | 37.5 | 34.7
  Month 9 : Very much better: number analyzed (Participants) | 16 | 122
  Month 9 : Very much better | 25.0 | 11.5
  Month 9 : Much better: number analyzed (Participants) | 16 | 122
  Month 9 : Much better | 50.0 | 50.8
  Month 9 : Somewhat better: number analyzed (Participants) | 16 | 122
  Month 9 : Somewhat better | 25.0 | 36.1
  Month 12 : Very much better: number analyzed (Participants) | 16 | 122
  Month 12 : Very much better | 25.0 | 13.9
  Month 12 : Much better: number analyzed (Participants) | 16 | 122
  Month 12 : Much better | 56.3 | 50.8
  Month 12 : Somewhat better: number analyzed (Participants) | 16 | 122
  Month 12 : Somewhat better | 18.8 | 31.1
  Month 18 : Very much better: number analyzed (Participants) | 16 | 118
  Month 18 : Very much better | 31.3 | 14.4
  Month 18 : Much better: number analyzed (Participants) | 16 | 118
  Month 18 : Much better | 43.8 | 47.5
  Month 18: Somewhat better: number analyzed (Participants) | 16 | 118
  Month 18: Somewhat better | 25.0 | 36.4
  Month 24 : Very much better: number analyzed (Participants) | 16 | 117
  Month 24 : Very much better | 18.8 | 15.4
  Month 24 : Much better: number analyzed (Participants) | 16 | 117
  Month 24 : Much better | 56.3 | 53.0
  Month 24 : Somewhat better: number analyzed (Participants) | 16 | 117
  Month 24 : Somewhat better | 25.0 | 29.1

13. Secondary Outcome: Percentage of Participants Agreeing That They Are Satisfied by the Treatment
Description: The subject's satisfaction with the procedure was assessed using a Subject Satisfaction Questionnaire. Question 7 was answered on a 4-grade scale: Overall, how satisfied are you with the treatment result? Very satisfied/ Satisfied/ Somewhat satisfied/ Not satisfied.
Time Frame: Treatment group: Months 6, 9, 12, 18 and 24
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Group A: Sculptra | Group B: Sculptra
Number analyzed (Participants) | 16 | 124
percentage of participants
  Month 6 : Somewhat satisfied | 6.3 | 19.4
  Month 6 : Satisfied | 43.8 | 49.2
  Month 6 : Very satisfied | 50.0 | 29.8
  Month 9 : Somewhat satisfied: number analyzed (Participants) | 16 | 122
  Month 9 : Somewhat satisfied | 12.5 | 22.1
  Month 9 : Satisfied: number analyzed (Participants) | 16 | 122
  Month 9 : Satisfied | 43.8 | 55.7
  Month 9: Very satisfied: number analyzed (Participants) | 16 | 122
  Month 9: Very satisfied | 43.8 | 19.7
  Month 12: Somewhat satisfied: number analyzed (Participants) | 16 | 122
  Month 12: Somewhat satisfied | 6.3 | 18.9
  Month 12 : Satisfied: number analyzed (Participants) | 16 | 122
  Month 12 : Satisfied | 37.5 | 53.3
  Month 12: Very satisfied: number analyzed (Participants) | 16 | 122
  Month 12: Very satisfied | 56.3 | 23.8
  Month 18: Somewhat satisfied: number analyzed (Participants) | 16 | 118
  Month 18: Somewhat satisfied | 6.3 | 20.3
  Month 18 : Satisfied: number analyzed (Participants) | 16 | 118
  Month 18 : Satisfied | 43.8 | 44.1
  Month 18: Very satisfied: number analyzed (Participants) | 16 | 118
  Month 18: Very satisfied | 50.0 | 33.1
  Month 24 : Somewhat satisfied: number analyzed (Participants) | 16 | 117
  Month 24 : Somewhat satisfied | 12.5 | 14.5
  Month 24 : Satisfied: number analyzed (Participants) | 16 | 117
  Month 24 : Satisfied | 37.5 | 54.7
  Month 24 : Very satisfied: number analyzed (Participants) | 16 | 117
  Month 24 : Very satisfied | 50.0 | 29.1

14. Secondary Outcome: Percentage of Participants Who Received Positive Feedback About Their Look From Family, Friends and Colleagues
Description: The subject's satisfaction with the procedure was assessed using a Subject Satisfaction Questionnaire. Question 8: Did you get any feedback about your look from your family, friends and colleagues? Positive/Negative/No feedback.
Time Frame: Treatment group: Months 6, 9, 12, 18 and 24
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Group A: Sculptra | Group B: Sculptra
Number analyzed (Participants) | 16 | 124
percentage of participants
  Month 6 | 81.3 | 71.0
  Month 9: number analyzed (Participants) | 16 | 122
  Month 9 | 81.3 | 68.9
  Month 12: number analyzed (Participants) | 16 | 122
  Month 12 | 81.3 | 77.9
  Month 18: number analyzed (Participants) | 16 | 118
  Month 18 | 87.5 | 75.4
  Month 24: number analyzed (Participants) | 16 | 117
  Month 24 | 93.8 | 76.1

15. Secondary Outcome: Percentage of Participants Who Recommended This Treatment to Their Friends
Description: The subject's satisfaction with the procedure was assessed using a Subject Satisfaction Questionnaire. Question 9 was a yes or no question: Would you recommend this treatment to friends?
Time Frame: Treatment group: Months 6, 9, 12, 18 and 24
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Group A: Sculptra | Group B: Sculptra
Number analyzed (Participants) | 16 | 124
percentage of participants
  Month 6 | 100.0 | 90.3
  Month 9: number analyzed (Participants) | 16 | 122
  Month 9 | 100.0 | 90.2
  Month 12: number analyzed (Participants) | 15 | 122
  Month 12 | 93.8 | 87.7
  Month 18: number analyzed (Participants) | 16 | 118
  Month 18 | 100.0 | 89.8
  Month 24: number analyzed (Participants) | 16 | 117
  Month 24 | 100.0 | 90.6

16. Secondary Outcome: Percentage of Participants Who Liked to Receive the Same Treatment Again
Description: The subject's satisfaction with the procedure was assessed using a Subject Satisfaction Questionnaire. Question 10 was a yes or no question: Would you like to receive the same treatment again?
Time Frame: Treatment group: Months 6, 9, 12, 18 and 24
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Group A: Sculptra | Group B: Sculptra
Number analyzed (Participants) | 16 | 124
percentage of participants
  Month 6: Yes | 100.0 | 85.5
  Month 9: Yes: number analyzed (Participants) | 16 | 122
  Month 9: Yes | 100.0 | 82.8
  Month 12 : Yes: number analyzed (Participants) | 16 | 122
  Month 12 : Yes | 93.8 | 83.6
  Month 18: Yes: number analyzed (Participants) | 16 | 118
  Month 18: Yes | 100.0 | 85.6
  Month 24 : Yes: number analyzed (Participants) | 16 | 117
  Month 24 : Yes | 93.8 | 86.3

ADVERSE EVENTS:
Time Frame: From start of study product administration up to 2 years 4 months
Description: Safety population included all participants in Group B who were treated with Sculptra or randomized to no-treatment group and participant in Group A who were treated with Sculptra.
Arm/Group | Group A: Sculptra | Group B: Sculptra | Group B: Control
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/124 | 0/63
Serious Adverse Events (participants affected / at risk) | 2/16 | 7/124 | 0/63
Other Adverse Events (participants affected / at risk) | 10/16 | 15/124 | 4/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Sculptra (N=16) | Group B: Sculptra (N=124) | Group B: Control (N=63)
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 — All SAEs were unrelated to the product and/or the injection procedure.
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 — All SAEs were unrelated to the product and/or the injection procedure.
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 — All SAEs were unrelated to the product and/or the injection procedure.
Removal of internal fixation (Surgical and medical procedures) | 0 | 1 | 0 — All SAEs were unrelated to the product and/or the injection procedure.
Basedow's disease (Surgical and medical procedures) | 0 | 1 | 0 — All SAEs were unrelated to the product and/or the injection procedure.
Gallbladder polyp (Hepatobiliary disorders) | 0 | 1 | 0 — All SAEs were unrelated to the product and/or the injection procedure.
Cardiac neoplasm unspecific (Cardiac disorders) | 0 | 1 | 0 — All SAEs were unrelated to the product and/or the injection procedure.
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 — All SAEs were unrelated to the product and/or the injection procedure.
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — All SAEs were unrelated to the product and/or the injection procedure.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Sculptra (N=16) | Group B: Sculptra (N=124) | Group B: Control (N=63)
Dental caries (Gastrointestinal disorders) | 0 | 8 | 1
Implant site nodule (General disorders) | 0 | 7 | 0
Arrhythmia (Cardiac disorders) | 2 | 0 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0
Xerophthalmia (Eye disorders) | 1 | 3 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 2
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 2 | 0
Asthenia (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 1 | 2 | 0
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 2 | 0
Influenza (Infections and infestations) | 1 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 5 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 10 | 4
Urinary tract infection (Infections and infestations) | 1 | 5 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 1
Calcium deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cervix disorder (Reproductive system and breast disorders) | 1 | 0 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 1 | 1 | 0
Menstrual disorder (Reproductive system and breast disorders) | 1 | 3 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Alopecia areata (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 5 | 2
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The initial publication of data from the Study must be a multi-center publication. Any subsequent publication/presentation must be sent to Sponsor for review 60 days before submission for publication/presentation to allow Sponsor to protect patentable inventions/confidential information. Site and Investigator agree to amend proposed publication/presentation, remove such confidential information from it, or postpone submission for a further 60 days/until intellectual property filings take place.

DOCUMENTS (2):
  • Study Protocol (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT04132518/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT04132518/SAP_001.pdf